CLINICAL TRIAL: NCT04804774
Title: Single-Arm Trial of a Virtual Weight Control Program Tailored for Adults With Type 2 Diabetes on Glycemic Control (VITAL)
Brief Title: Virtual Weight Control Program Tailored for Adults With Type 2 Diabetes (VITAL)
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor - Clinical Nutrition and Metabolism, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC2021-014
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Type2 Diabetes; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WW program modified for people with Type 2 diabetes (Experimental): Includes weekly Virtual Workshops and use of the WW App.
  Interventions: Behavioral: WW program modified for people with Type 2 diabetes

INTERVENTIONS:
Behavioral: WW program modified for people with Type 2 diabetes — This 6-month intervention includes the use of WW's mobile app, weekly virtual workshops, and private online community. The program involves: self-monitoring of weight, dietary intake, and physical activity; dietary changes; increasing physical activity; shift in mindset; and behavioral strategies to manage goals. Participants will set goals and weigh-in with a coach via virtual workshop weekly and be encouraged to use the app and private online community daily. The virtual workshop features a behavior change technique and enables the participant to practice it to support their goals. Participants are given a personalized food plan based on expert healthy eating guidelines, an activity plan to promote regular physical activity and techniques to help shift mindset for lasting change. The coach will help with goal setting, overcoming setbacks, and follow-up on progress toward goals weekly. Participants will be encouraged to participate in a private Facebook group for motivational support.

SUMMARY:
The purpose of the study is to evaluate the effect of the WW program on people with Type 2 diabetes and the effect on glycemic control. This study will be a 6 month prospective, single arm clinical trial coordinated by Pennington Biomedical Research Center. Up to 150 participants will be recruited across 3 sites. Participants will have Type 2 diabetes and overweight/obesity.

DETAILED DESCRIPTION:
While weight loss (2-5% of total bodyweight) with clinical interventions has been shown to improve glycemic control in patients with Type II Diabetes clinic-based interventions are costly and have poor accessibility for the majority of patients. Commercial weight loss programs like WW (formerly Weight Watchers) are more affordable and accessible than clinic-based modalities, and have been shown to produce effective weight loss in adults with additional improvements in glycemic control. A randomized trial of a modified WW program for patients with Type II Diabetes showed significant reductions in weight and improved glycemic control (HbA1c) compared to standard of care diabetes nutrition counseling and education. Here, we extend prior work by leveraging the efficacy of the WW program for Type II Diabetes, virtually, to increase its reach and its impact on glycemic control. This study aims to test a novel, web-based weight loss intervention from one of the largest and most evidence-based proprietary weight loss programs in the world.

Intervention will consist of the WW program modified for people with Type 2 diabetes including weekly Virtual Workshops and use of the WW App. Primary outcomes are any change in HbA1c% over the 6-month intervention. Secondary endpoints are any change in HbA1c% at 3 months, as well as changes at 3 and 6 months in weight, Diabetes Distress Scale, Impact of Weight on Quality of Life, Pittsburgh Sleep Quality Index, hypoglycemic events, WHO-5 Well-being Index, and diabetes medication changes.

ELIGIBILITY:
Inclusion Criteria:

- 1. Participant reported diagnosis of Type 2 diabetes 2. HbA1c between 7%-11% (inclusive) 3. BMI 27-50 kg/m2 (inclusive) 4. Age range - 18 - 70 years (inclusive) 5. On stable regimen of all medications (including diabetes) for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted) 6. Willingness to attend weekly WW Virtual Workshops and to participate in WW Digital program 7. Access to a iOS smart phone device with internet 8. Willing to follow all requirements of study protocol including blood draws at baseline, week 12, and week 24.

9. Willing and able to provide a valid email address for use in the study 10. Must be able to communicate (oral and written) in English 11. Under the care of a physician who will be responsible for managing the subject's diabetes and a subject who is willing to give release to provide their treating MD with information about the trial

Exclusion Criteria:

* 1. Participation in a weight control program within the past 3 months 2. Weight loss of ≥ 5 kg in the previous 6 months 3. Taking prescription or OTC weight loss medications within last 4 weeks 4. History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve) 5. History of major surgery within three months of enrollment 6. Currently taking other medications that affect weight (e.g., paroxetine, tricyclics, anti-psychotics) 7. Type 1 diabetes 8. Those on insulin or insulin secretagogues 9. Renal insufficiency consisting of potassium over 5.5 (mmol/L) on a non-hemolyzed specimen, or a creatinine over 2.5 mg/dL 10. Bilirubin over 3 (mg/dL) or an albumin less than 3 (g/dL) 11. ALT > 3 (IU/L) times the upper limit of normal (normal range is 7-56) 12. Evidence of more than 1 severe hypoglycemic event (episode requiring emergency medical services) in the past 12 months, unless the participant's treating physician provides written clearance for participation.

  13. Hemoglobinopathy that interferes with measurement of hemoglobin A1c 14. Those on higher doses of diuretics (furosemide 40mg or higher or comparable) 15. Unstable heart disease (an ongoing workup or treatment for a cardiac symptom such as unstable angina, coronary ischemia) 16. Presence of implanted cardiac defibrillator 17. Blood pressure ≥180/100 mm Hg. If a potential participant has a BP above the inclusion criteria it is acceptable to re-test this potential participant within one week of the original test.

  18. Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 months. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable 19. Orthopedic limitations that would interfere with ability to engage in regular physical activity 20. Uncontrolled gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease 21. Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Persons with successfully resected non-melanoma carcinoma of the skin may be enrolled.

  22. Dementia, psychiatric illness, or substance abuse that may interfere with adherence (e.g. illness that is currently unstable or resistant to first-line therapy; substance abuse in the past year), 23. History within the past five years of clinically diagnosed eating disorders including anorexia nervosa or bulimia nervosa.

  24. Women who are pregnant, lactating, trying to become pregnant or unwilling to use an effective means of birth control 25. Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and unwilling to limit intake to less than 3 drinks per drinking day during study participation 26. Participation in another clinical trial within 30 days prior to enrollment. 27. Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Change in % HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center; Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealth University; Stephen Anton, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Pennington Biomedical Research, Baton Rouge, Louisiana
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No